CLINICAL TRIAL: NCT01933633
Title: Study of Pregnancy Rate After Exercise Training Prior to Assisted Fertilisation in Overweight/Obese Women
Brief Title: Improved Fertility After Exercise in Overweight/Obese Women
Acronym: FertilEX
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment proceeded to slowly
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Alesund Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FertilEX
Record Dates: First submitted 2013-08-28; First posted 2013-09-02 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Obesity; Infertility, Female
Keywords: Pregnancy; Fertility; exercise; Fertilization in vitro
MeSH Terms: conditions — Obesity; Infertility, Female; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Regular exercise training for 10 weeks prior to assisted fertilisation
  Interventions: Behavioral: Exercise
- Control (No Intervention): Standard care

INTERVENTIONS:
Behavioral: Exercise
  Arms: Exercise

SUMMARY:
Overweight/obesity is associated with sub-fertility. The investigators will assess if regular exercise training prior to assisted fertilization will improve pregnancy rate in overweight/obese women referred to assisted fertilization. It is expected that training will be successful in increasing pregnancy rate

DETAILED DESCRIPTION:
Obesity is associated with several diseases, as type 2 diabetes, cardiovascular disease and some types of cancer, this is of great concern for the public health. Also, of more immediate importance for these women; obesity is associated with increased risks of sub-fertility. The overall aim of the current project is to expand the knowledge about effective interventions to prevent the increasing prevalence of obesity-associated sub-fertility in population.

One cause of the increased referral rate for in-vitro fertilization is the growing prevalence of overweight and obesity. Currently, about 700 couples are annually referred for in-vitro fertilization at St.Olav's Hospital. In this interdisciplinary trial, involving physiotherapists, exercise physiologists, gynecologists, and basic researchers, the effects of regular high intensity exercise training on fertility in sub-fertile overweight and obese women will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (weight in kg/height in cm squared) >25
* accepted for assisted fertilization treatment at St.Olav's hospital

Exclusion Criteria:

* low responders, defined as AMH <2 pmol/L or < 5 oocytes in prior in vitro fertilisation (IVF)/Intracytoplasmic sperm injection (ICSI) cycles or antral follicle count (AFC) < 5
* current or previous Metformin use (a wash-out period of > four weeks)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | 7 weeks after assisted fertilisation
  The primary outcome measure is ongoing pregnancy, defined as the sonographic evidence of intrauterine gestational sac and fetal heart activity at seven weeks of gestation.

CONTACTS AND LOCATIONS:
Overall Officials: Trine Moholdt, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (2):
- Norway (2):
  - Ålesund Hospital, Ålesund
  - St Olavs Hospital, Trondheim

REFERENCES:
- [Background] Lundgren KM, Romundstad LB, von During V, Morkved S, Kjotrod S, Moholdt T. Exercise prior to assisted fertilization in overweight and obese women (FertilEX): study protocol for a randomized controlled trial. Trials. 2016 Jun 1;17(1):268. doi: 10.1186/s13063-016-1398-x. PMID 27250851
- [Result] Kiel IA, Lundgren KM, Morkved S, Kjotrod SB, Salvesen O, Romundstad LB, Moholdt T. Women undergoing assisted fertilisation and high-intensity interval training: a pilot randomised controlled trial. BMJ Open Sport Exerc Med. 2018 Jul 17;4(1):e000387. doi: 10.1136/bmjsem-2018-000387. eCollection 2018. PMID 30057778